CLINICAL TRIAL: NCT06386874
Title: The Efficacy of a Frequency-tuned Electromagnetic Field Treatment in Facilitating the Recovery of Subacute Ischemic Stroke Patients - a Pivotal Study (the "EMAGINE 2.0" Study)
Brief Title: EMAGINE 2.0 - Electromagnetic Field Ischemic Stroke - Novel Subacute Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrainQ Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BQ7
Record Dates: First submitted 2024-04-16; First posted 2024-04-26 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: subjects will be assigned (1:1 allocation ratio) to either active or sham study intervention using the BQ3. system
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study, Sponsor, subjects and Investigators will be blinded to the device setting (Active/Sham). The study site team members receiving, storing, dispensing, preparing, and administering the study interventions will be blinded (except the unblinded randomizer). Subjects' caregivers will also be blinded. There are no differences in the active and sham device appearance. Due to the non-invasive nature of the treatment, as well as the physical characteristic of the EMF, there is no noticeable difference between sessions conducted using an active or a sham device, facilitating full blinding of both subjects and Investigators.
  An independent unblinded statistician (not the study statistician) will perform the assessments described. Only the unblinded statistician and members of the DSMB will be exposed to the interim report.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BQ 3.0 Sham Stimulation Group (Sham Comparator): Q Therapeutic System (BQ 3.0) sham stimulation group:
  Device used: Q Therapeutic System (BQ 3.0)
  In Stage 1: 45 sessions over a period of 9 weeks (5 treatments per week) of sham study intervention with BQ 3.0 (frequency and intensity parameters will be set to zero so that no stimulation is delivered) including a standardized, pre-defined and evidence-based physical and occupational therapy regimen concurrent with the study intervention.
  Interventions: Device: Q Therapeutic System (BQ 3.0) - Sham; Device: Q Therapeutic System (BQ 3.0) - Active
- BQ 3.0 Active Stimulation Group (Active Comparator): Q Therapeutic System (BQ 3.0) active stimulation group:
  Device used: Q Therapeutic System (BQ 3.0)
  In Stage 1: 45 sessions over a period of 9 weeks (5 treatments per week) of active study intervention with the BQ 3.0 (frequency and intensity parameters will be set to 1-100 Hz.; 0.1-1.0 G), including a standardized, pre-defined and evidence-based physical and occupational therapy regimen concurrent with the study intervention.
  Interventions: Device: Q Therapeutic System (BQ 3.0) - Sham; Device: Q Therapeutic System (BQ 3.0) - Active

INTERVENTIONS:
Device: Q Therapeutic System (BQ 3.0) - Sham — The BQ 3.0 is a medical device that produces and delivers non-invasive, extremely low intensity and frequency (1-100 Hz.; 0.1-1.0 G), frequency tuned electromagnetic fields in order to stimulate neuronal networks with the aim of reducing disability and promoting neurorecovery. Frequency and intensity parameters will be set to zero so that no stimulation is delivered.
  Other Names: BQ 3.0 Sham Stimulation Group
Device: Q Therapeutic System (BQ 3.0) - Active — The BQ 3.0 is a medical device that produces and delivers non-invasive, extremely low intensity and frequency (1-100 Hz.; 0.1-1.0 G), frequency tuned electromagnetic fields in order to stimulate neuronal networks with the aim of reducing disability and promoting neurorecovery
  Other Names: BQ 3.0 Active Stimulation Group Interventions

SUMMARY:
This is a multicenter study that will be conducted at approximately 20 centers and up to 30 centers, if the sample size will be increased following interim assessment.

The Q Therapeutic System (BQ 3.0) is a wearable medical device that produces and delivers non-invasive, extremely-low-intensity and low-frequency, frequency-tuned electromagnetic fields in order to stimulate neuronal networks with the aim of reducing disability and promoting neurorecovery.

The Q Therapeutic System (BQ 3.0) is indicated for adjunctive use in a clinical facility or home setting, in addition to standard-of-care therapies.

* In Stage 1 (starting 4-21 days after the index stroke event to day 90 post stroke), participants will be randomly assigned (1:1) to receive either active or the sham treatments, up to 5 times a week, and at least to a total of 45 treatments.
* In Stage 2 (day 90 to day 180 post stroke), participants in both the active and the control group will be allowed to continue to receive active treatments, up to 5 times per week.
* In stage 3 (day 180 to day 270 post stroke), participants will not receive any treatments and would be followed up until the final visit at day 270.

Each session will last approximately 60 minutes, with stimulation activated for up to 40 minutes, in conjunction with a home-based exercise program. Treatments may be administered in the hospital, in the clinic or in a home setting.

The study will enroll 100-122 adult subjects who will be randomly assigned (1:1 allocation ratio) to either active or sham study intervention using the BQ 3.0 system.

DETAILED DESCRIPTION:
The study intervention will be initiated 4-21 days after the index stroke event and will consist of 5 treatments per week until the primary endpoint follow-up visit, at day 90 (±15) after the onset of the index stroke. A minimum of 45 treatment sessions should be completed during this stage, with a potential of a maximum of 72 treatment sessions, depending on the start date of the first treatment and the timing of the 90-day follow-up visit. Though, participants and sites will be guided to conduct the 90 days follow-up visit as soon as possible after the 45th treatment session and within up to 7 days from the 45th treatment and after the window opening.

Each treatment session will last approximately 60 minutes and include 40 minutes of active or sham stimulation. Subjects in both groups will be asked to perform a home-based exercise program for the upper and the lower limb, concurrent with the study intervention.

Screening phase:

Prospective subjects, who are 3 to 21 days post-stroke, may be offered informed consent to participate in the study at either:

a participating inpatient or outpatient center, non-participating inpatient or outpatient center, in accordance with both the participating and the non-participating centers' policy, or home Consented subjects, who are 4 to 21 days post-stroke, will be screened for eligibility to participate in the treatment phase of the study.

Eligible subjects will be randomly assigned, at a 1:1 allocation ratio, to either the active or sham study intervention groups.

Stimulation with the Q Therapeutic System (BQ 3.0) does not produce any noticeable sound, light, or tactile sensation which could disclose the treatment arm assignment, making this device ideal for testing in a sham-controlled design. During sham treatment sessions, for purposes of maintaining the blind, the device will function as if it is delivering the therapy (i.e., the device will turn on and all indicators will function), but the frequency and intensity parameters, which are not visible to the subject or site study members (or any blinded personnel), will be set to zero so that no stimulation is delivered.

Stage 1 (day 4 to day 90 (±15) post-stroke) - double-blind sham-controlled:

Efforts should be made to initiate the 1st treatment as early as possible within the window of recruitment, and target to complete a first treatment within 6 days from admission to a participating IRF (where applicable). The study intervention will be initiated 4-21 days after the index stroke event and will consist of 5 treatments per week until the primary endpoint follow-up visit, at day 90 (±15) after the onset of the index stroke. Each treatment session will last approximately 60 minutes and include 40 minutes of active or sham stimulation. Subjects in both groups will be asked to perform a home- based exercise program for the upper and the lower limb, concurrent with the study intervention. The program will be standardized, pre-defined, home-based, and aligned with standard-of-care1.

The participant and their caregiver will be trained on the use of the device and exercise program. Treatment sessions will be completed by the subject with the assistance of a trained caregiver, as needed. Periodic supervision will be provided by the study team (combined audio and video remote conferencing or audio only, if video is not available). A sponsor's representative may provide in-person or remote technical support to the participant and their caregiver, as well as device training, as needed.

Subjects will undergo a detailed interim outcome assessment on the 45th (±4) day after the onset of the index stroke, and a detailed primary endpoint outcome assessment on the 90th (±15) day after the onset of the index stroke. In addition, a focused, long-term outcome assessment on the 180th (±15) day after the onset of the index stroke will be performed.

Stage 2 (day 90 (±15) to day 180 (±15) post-stroke) - open-label:

Subjects in both the active and the sham groups (active /sham), who were adherent to the treatment in Stage 1 (defined as at least 35 completed treatment sessions in Stage 1) will be allowed to continue to receive active EMFstimulation treatments (i.e., with the electromagnetic therapy turned on).

Up to 5 active treatments per week will be completed, starting following the primary endpoint assessment follow-up visit at 90 (±15) days after the onset of the index stroke and continuing until the follow-up visit at 180 (±15) days after the onset of the index. Technically, a maximum of 86 treatment sessions can be completed during stage 2, depending on the timing of the 90-day and 180-day follow-up visits.

The blind, with respect to the group allocation in Stage 1, would be maintained for all parties (participants, investigators, assessors and Sponsor) until the trial completion and database lock.

Each session will last approximately 60 minutes and include 40 minutes of active stimulation. Subjects will be asked to perform a home-based exercise program, concurrent with the study intervention.

Treatment sessions will be completed by the subject with the assistance of a trained caregiver, as needed. Periodic supervision will be provided by the study team (combined audio and video remote conferencing or audio only, if video is not available). A sponsor's representative willmay provide in-person or remote technical support to the participant and their caregiver, as well as device training, as needed.

All subjects, including those who decided not to continue to receive treatments in Stage 2, will undergo a detailed follow-up assessment on the 180th (±15) day after the onset of the index stroke.

Stage 3 (day 180 (±15) to day 270 (±15) post-stroke):

At this Stage, no treatments sessions will take place. All subjects, including those who decided not to continue to receive treatments in Stage 2, will undergo In addition, aa focused, long-term outcome assessment on the 180th 270th (±15) day after the onset of the index stroke will be performed.

Any adverse events and device deficiencies occurring during the period of subject's participation in the trial will be recorded.

Participation in the study will not replace any of the usual care patient should receive.

ELIGIBILITY:
Inclusion Criteria:

1. mRS score of 3 or 4.
2. FMA-UE score between 10-45 (inclusive) of impaired limb.
3. SAFE score >0.
4. Age 22 to 80 years of age (inclusive).
5. Diagnosed with an ischemic stroke, confirmed by CT4 or MRI5 imaging.
6. First ever ischemic stroke, or a recurring ischemic stroke6 occurring at least 3 months after the previous stroke (any stroke), without residual neurological impairment or disability before current stroke.
7. Four to 21 days from stroke onset (or last known well).
8. Pre-stroke mRS of 0.
9. Able to sit with the investigational device for 40 consecutive minutes, in the opinion of the investigator or designee.
10. Can follow a 3-step command, such as "take the paper, fold it in half, and return it to me".
11. Willingness to participate in an exercise activity during study intervention sessions.
12. Availability of a relative or other caregiver able to assist in operating an application installed on a mobile device, including a video call, and assist the participant with the exercising program.
13. If female, not pregnant (as confirmed by a urine or a blood test, or as determined by an official medical document) or breastfeeding and with no ability to become pregnant or on an acceptable method of contraception during the study
14. Informed consent signed by subject.

Exclusion Criteria:

1. Hemineglect impairment (NIHSS item 11, score >0).
2. Implanted active electronic or passive MR-incompatible devices.
3. Pre-existing major neurological condition (eg, Alzheimer's disease, Parkinson's disease, multiple sclerosis, traumatic brain injury, spinal cord injury) or pre-existing physical limitation that would interfere significantly with the subject's participation in the study and/or confound neurological or functional evaluation.
4. Active epilepsy or currently taking anti-epileptic medication (indicated for the treatment of a seizure disorder), or any epileptic seizure in the last 5 years
5. Significant visual disturbances, pre-existing or resulting from the index stroke, that cannot be corrected and that would interfere significantly with the subject's participation in the study and/or confound neurological or functional evaluation.
6. Unstable serious illness/condition (eg, active cancer, severe heart failure, active major psychiatric condition) or life expectancy of less than 12 months.
7. A known severe allergic reaction to acrylic-based adhesives.
8. Alcohol abuse and/or illicit drug abuse in the past 6 months, which is likely to influence ability to fully participate in the trial.
9. Participation in another trial that would conflict with the current study or clinical endpoint interference may occur.
10. Employee of the Sponsor.
11. Prisoner.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Modified Rankin Scale | 4 to 21 days following an ischemic stroke to 90-day post-stroke
  Proportion of subjects achieving an excellent outcome defined as a Modified Rankin Scale (mRS) score of 0-1 at the 90-day post-stroke assessment, reflecting freedom from disability.

SECONDARY OUTCOMES:
Ordinal shift analysis of the mRS (trichotomized at 0-1, 2, 3-6) (Key Secondary Effectiveness Endpoint) | baseline to the 90-day post-stroke assessment
Change from Baseline in Modified Rankin Scale (Key Secondary Effectiveness Endpoint) | baseline (4-21 days post-stroke) to 90 days post-stroke
  To show that the BQ therapy is effective in reducing disability levels
Proportion of subjects achieving functional independence (mRS score of 0-2) (Key Secondary Effectiveness Endpoint) | at the 90-day post-stroke assessment
  To show that the BQ therapy is effective in achieving functional independence.
Stroke Impact Scale Hand Domain (Lead Secondary Endpoint) | baseline (4 to 21 days following an ischemic stroke) to 90-day post-stroke
  Patient reported hand function - To show that the BQ therapy is effective in improving upper limb impairment and function
Stroke Impact Scale 16 | baseline (4 to 21 days following an ischemic stroke) to 90-day post-stroke
  Patient-reported physical function - To show that the BQ therapy is effective in improving physical function
10-meter Walk Test | change from baseline to 90 days post-stroke
  The Functional Ambulation Categories (FAC) will be collected concurrent to the 10MWT to assess the level of independent ambulation.
Box and Block Test | baseline (4 to 21 days following an ischemic stroke) to 90-day post-stroke
  Arm motor function - To show that the BQ therapy is effective in improving Arm motor function
Evaluation of 5-level EQ-5D | At 90-days post-stroke
  Health-related quality of life - To show that the BQ therapy is effective in achieving health-related quality of life (HRQoL)
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | baseline (4 to 21 days following an ischemic stroke) to 90-day post-stroke
  upper limb impairment - To show that the BQ therapy is effective in achieving reducing upper limb impairment, and improving upper limb function
Nine-Hole Peg Test | change from baseline to 90-days post-stroke
  finger dexterity - To show that the BQ therapy is effective in achieving reducing upper limb impairment, and improving upper limb function
The proportion of subjects within those in the active group who continued to receive treatments in Stage 2, achieving an excellent outcome (defined as a mRS of 0-1) at the 180-day post-stroke assessment. | at the 180-day post-stroke assessment
  To show, within those in the active group who continued to receive treatments in Stage 2, that the BQ therapy is effective in attaining freedom from disability, as well as reducing global disability, at 6 months post-stroke in disabled patients when initiated 4 to 21 days following an ischemic stroke.
The proportion of patients within those in the active group who continued to receive treatments in Stage 2, who achieved an excellent outcome defined as a mRS score of 0-1 at the 90-day post-stroke assessment and had an mRS >1 at 180-day post-stroke | at 180 days post-stroke
  To show, within those in the active group who continued to receive treatments in Stage 2, that the BQ therapy is effective in attaining freedom from disability, as well as reducing global disability, at 6 months post-stroke in disabled patients when initiated 4 to 21 days following an ischemic stroke
The proportion of patients within those in the active group who continued to receive treatments in Stage 2, who achieved an excellent outcome defined as mRS score of 0-1 at the 180-day post-stroke assessment and had an mRS >1 at 270 days post-stroke. | at 270 days post-stroke
  To show, within those in the active group who continued to receive treatments in Stage 2, that the effect attained in obtaining freedom from disability, as well as reducing global disability, is maintained at 6- and 9- months post-stroke in disabled patients with upper limb motor impairment when initiated 4 to 21 days following an ischemic stroke.
Ordinal shift analysis of the mRS (4 levels at 0, 1, 2, 3-6) from the 90-day post-stroke assessment to 180-day post-stroke assessment, within those in the active group who continued to receive treatments in Stage 2 | from the 90-day post-stroke assessment to 180-day post-stroke assessment
The proportion of patients who improved by at least 1 level on the mRS from the 90-day post-stroke assessment to 180-day post-stroke assessment, within those in the active group who continued to receive treatments in Stage 2. | from the 90-day post-stroke assessment to 180-day post-stroke assessment
  To show, within those in the active group who continued to receive treatments in Stage 2, that the BQ therapy is effective in attaining freedom from disability, as well as reducing global disability, at 6 months post-stroke in disabled patients when initiated 4 to 21 days following an ischemic stroke
The proportion of subjects within those in the sham group who continued to receive treatments in Stage 2, achieving an excellent outcome (defined as a mRS of 0-1) at the 180-day post-stroke assessment, and had an mRS >1 at 90 days post-stroke. | from the 90-day assessment to the 180-day assessment
  To show, within those in the sham group who continued to receive treatments in Stage 2 that the BQ therapy is effective in attaining freedom from disability, as well as reducing global disability, at 6 months post-stroke in disabled patients when initiated 90 days following an ischemic stroke

OTHER OUTCOMES:
Serious procedure or device related adverse events & device deficiencies | Through study completion, an average of 90 ± 15 days post-stroke
  To characterize the safety profile of the BQ therapy and to show that the BQ 3.0 performs reliably.
Change in Montreal Cognitive Assessment (global cognitive function) | at 90-day post-stroke
  To show that the BQ therapy is effective in reducing cognitive impairment, at 3 months post-stroke, when initiated 4 to 21 days following an ischemic stroke.
Change in Patient Health Questionnaire-8 (depression) | at 90-day post stroke
  To show that the BQ therapy is effective in reducing depression, at 3 months post-stroke, when initiated 4 to 21 days following an ischemic stroke.
Academic Medical Center Linear Disability Scale (granular level of disability) | At 90 days post stroke
  To show that the BQ therapy is effective in reducing fine-grained level of disability at 3 months post-stroke
Proportion of subjects achieving functional independence (modified Rankin Scale score of 0-1) | at 45 days post-stroke
  To show that the BQ therapy is effective in increasing functional independence at 1.5 months post-stroke
Zarit Burden Interview | at midterm, 90 days post-stroke, 180 days post-stroke, and 270 days post-stroke.
  To formally evaluate the cost-effectiveness of the BQ therapy via caregiver burden.
Formal cost-effectiveness analysis over a lifetime horizon from the perspective of the United States healthcare system. | will be assessed at MidTerm (45 Day ± 4 days post- stroke) , Day-90 and D-180 post stroke
  To formally evaluate the cost-effectiveness of the BQ therapy over a lifetime horizon from the perspective of the United States healthcare system
Relationship between adherence to treatment as measured by the Qompass and the clinical outcomes. | Will be assessed upon data base lock
  To explore the relationship between adherence to treatment as measured by the Qompass and clinical outcomes.
The proportion of patients within those in the sham group who continued to receive treatments in Stage 2 who improved from the 90-day assessment to 180-day and the improvement was maintained at 270 days post-stroke | At 180 days post stroke and 270 days post-stroke
  To show, within those in the sham group who continued to receive treatments in Stage 2 that the BQ therapy is effective in improving functional independence at 6 months post-stroke, when initiated 90 days following an ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Saver, MD, Study Chair — Coordinating PI; Joel Stein, MD, Principal Investigator — Coordinating PI
Locations (14):
- United States (14):
  - Rancho Research Institute, Downey, California
  - MedStar National Rehabililtaion Hospital,, Washington D.C., District of Columbia
  - Brooks Rehabilitation Hospital, Jacksonville, Florida
  - Emory University School of Medicine, Altanta, Georgia
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - KUMC- KU Medical Center, Kansas City, Kansas
  - Hackensack Meridian JFK Johnson Rehabilitation Institute, Edison, New Jersey
  - Kessler Foundation for Rehabilitation, West Orange, New Jersey
  - New York-Presbyterian Brooklyn Methodist Hospital Inpatient Rehabilitation Unit, Brooklyn, New York
  - Burke Rehabilitation Hospital, White Plains, New York
  - Atrium Health Carolinas Rehabilitation, Charlotte, North Carolina
  - Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania
  - UTHealth Houston, Houston, Texas
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
will be shared following site level approval